CLINICAL TRIAL: NCT04350905
Title: Characterization of Skin Immunity to Aedes Aegypti Saliva in Dengue-Endemic Participants in Cambodia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 999920053; 20-I-N053
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2021-04-09

CONDITIONS: Vector Borne Diseases
Keywords: Vector-Borne Diseases; Immune Response; Mosquito Feeding; Arbovirus; Southeast Asia
MeSH Terms: conditions — Vector Borne Diseases

STUDY DESIGN:
Intervention Model Description: Participants were all exposed to 5 uninfected Aedes aegypti mosquitos on their forearm. Biopsies were taken of bitten and unbitten skin.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mosquito Feeding (Experimental): Each participant will receive one mosquito feeding with 5 starved female Aedes aegypti mosquitoes.
  Interventions: Other: Mosquito Feeding

INTERVENTIONS:
Other: Mosquito Feeding — Mosquito feedings will be conducted with Aedes aegypti colonies raised at the CNM (National Malaria Center) Malaria and Vector Research Laboratory (MVRL), an established state of the art insectaries for mosquitoes was built in 2014 to ACL2 (arthropodcontainment level 2)-level specifications.

SUMMARY:
Background:

Mosquito-borne viruses like dengue cause major illness and death worldwide, particularly in Southeast Asia. When mosquitoes deliver a virus into the skin of humans, they also leave saliva. Researchers want to learn more about skin immunity to mosquito saliva. They hope this will help with future vaccines and treatments for these diseases.

Objective:

To compare the early and late innate immune response in the skin of Aedes aegypti bitten versus unbitten skin.

Eligibility:

Healthy people ages 18-45 who live within about 15 km of the study site in Chbar Mon

Design:

Participants will have 3 visits.

The baseline/screening visit will include:

Medical and medication history

Questions about participants demographic information, mosquito biting risk factors, and responses to mosquito or other insect bites

Physical exam

Urine sample for some participants

Mosquito feeding. A feeding device will be placed on the participant s arm for up to 20 minutes. The insects will feed through a mesh on the bottom of the feeding device. Participants may be given standard treatments for any skin reactions.

Blood tests

Four skin biopsies taken from bitten and unbitten skin. Local anesthetic will be administered, and a small tool will be used to remove the participant s skin.

Participants will have a second visit the next day. They will have a physical exam and blood tests. They will have 1 skin biopsy.

Participants will have a final visit about 2 weeks later. They will have a physical exam and blood tests.

During the study, participants will be asked to take measures to prevent more mosquito bites.

DETAILED DESCRIPTION:
Mosquito-borne viruses continue to cause significant global morbidity and mortality, particularly in Southeast Asia. When mosquitoes deliver the virus into the skin of humans while probing for a blood meal, they deposit also saliva, which contains a myriad of pharmacologically active compounds that modulate the host immune system. Little is known about skin immunity to mosquito saliva, particularly in endemic volunteers as most clinical studies are performed in na(SqrRoot) ve individuals who have never or rarely been exposed to a particular mosquito vector. People living in endemic areas have had long-term repeated exposure to these vectors and therefore have different immune response to mosquito saliva, which could interfere with mosquito-borne disease vaccine effectiveness. Characterization of skin immunity via various technical modalities will be important in order to identify critical aspects of the innate and adaptive immune responses after a vector bite.

Here, we will execute a paired study of exposed-unexposed skin to carefully examine the innate and adaptive immune responses in the skin and blood to exposure of the saliva of Aedes aegypti, the mosquito vector of dengue, Zika, and chikungunya viruses. We will enroll 42 participants to undergo vector feeding and give blood samples at baseline and 2 and 14 days later. Additionally, participants will give skin punch biopsy samples of bitten (exposed) and unbitten (unexposed) skin. For analysis, we will group 10-12 participants in each of 4 technical modality cohorts or groups : 1) immunohistochemistry, 2) RNA sequencing, 3) flow cytometry, and 4) T-cell receptor sequencing. With the current rise of vector-borne diseases in the United States and around the world, we hope the results of this study contribute to future vaccine design and clinical development strategies for vector#borne diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

-Provision of signed and dated informed consent form

* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 - 45 years
* Live within approximately 15 km of study site
* In good general health as evidenced by medical history
* Willing to allow biological samples to be stored for future research.
* A female is eligible for this study if she meets 1 of the following:

  * Of non-childbearing potential (i.e., women who have had a hysterectomy or tubal

ligation or are postmenopausal, as defined by no menses in >=1 year).

--Of childbearing potential but has negative urine pregnancy test on Day 0

* Agrees to not use scented lotions, deodorants, or topical creams on each feeding day.
* Agrees to not take aspirin or any other NSAID (ex. ibuprofen) within 7 days of a biopsy.
* Agrees to not use oral or topical antihistamines or steroid creams or ointments throughout the

study without prior permission of Principal Investigator (PI).

EXCLUSION CRITERIA:

-Any underlying or current medical condition that, in the opinion of the investigator, would

interfere with participation in the study.

-History of severe allergic reaction (including to mosquito or other insect bites) with generalized

urticaria, angioedema, anaphylaxis, anaphylactoid reaction or any other reaction described by

the participant and deemed severe by the PI.

* Self-reported or known history of alcoholism or drug abuse within 6 months prior to enrollment
* Self-reported or known history of psychiatric or psychological issues that require treatment and

are deemed by the PI to be a contraindication to protocol participation.

-Any use of medications that affect blood clotting within 3 months or history of abnormal blood

clotting

-History of significant scarring such as keloids after previous biopsies, lacerations, abrasions,

surgeries, or other skin procedures (e.g., cosmetic piercings) that are deemed by the PI to be a

contraindication to protocol participation.

-Pregnant or breastfeeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Manning, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Kampong Speu Referral Hoispital, Chbar Mon, Cambodia

REFERENCES:
- [Background] Durnez L, Mao S, Denis L, Roelants P, Sochantha T, Coosemans M. Outdoor malaria transmission in forested villages of Cambodia. Malar J. 2013 Sep 17;12:329. doi: 10.1186/1475-2875-12-329. PMID 24044424
- [Background] Manning JE, Morens DM, Kamhawi S, Valenzuela JG, Memoli M. Mosquito Saliva: The Hope for a Universal Arbovirus Vaccine? J Infect Dis. 2018 Jun 5;218(1):7-15. doi: 10.1093/infdis/jiy179. PMID 29617849
- [Background] Huy R, Buchy P, Conan A, Ngan C, Ong S, Ali R, Duong V, Yit S, Ung S, Te V, Chroeung N, Pheaktra NC, Uok V, Vong S. National dengue surveillance in Cambodia 1980-2008: epidemiological and virological trends and the impact of vector control. Bull World Health Organ. 2010 Sep 1;88(9):650-7. doi: 10.2471/BLT.09.073908. Epub 2010 Apr 7. PMID 20865069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mosquito Feeding
Started | 42
Completed | 41
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mosquito Feeding
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Cambodia | 42
Exposure to Dengue [Count of Participants; unit: Participants] | 42

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Change in Early and Late Innate Immune Responses Using Gene Expression and Flow Cytometry in Participants' Skin
Description: Measurement of changes in the early and late innate immune response and cellular recruitment in bitten skin versus unbitten skin by: a) immunohistochemistry of target proteins at Day 0 timepoints b) immunophenotyping of innate immune cell subsets in dissociated skin sample at Day 0 timepoints c) determination of cytokine profile in dissociated skin sample supernatant at Day 0 timepoints d) differential cDNA expression prepared from skin RNA and analyzed via RNASeq at Day 0 timepoints
Time Frame: Day 0 timepoints
Population: Flow and RNAseq populations
Measure: Median (Inter-Quartile Range); unit: % of total dendritic cells
Arm/Group | Mosquito Feeding
Number analyzed (Participants) | 30
% of total dendritic cells
  % total DCs at 30 min | 50 [45 to 55]
  % activated dermal DCs at 30 min | 5 [3 to 8]

2. Primary Outcome: Measurement of Changes in the Adaptive Immune Response and Cellular Recruitment in the Skin of Bitten Versus Unbitten Skin After Sixth and Final Feeding in Each Vector Group.
Description: Measurement of changes in the adaptive immune response and cellular recruitment in bitten skin versus unbitten skin by: a) immunohistochemistry of target proteins at Day 2 timepoints b) phenotyping of adaptive immune cell subsets in dissociated skin sample at Day 2 timepoints c) determination of cytokine profile in dissociated skin sample supernatant at Day 2 timepoints d) differential cDNA expression prepared from skin RNA and analyzed via RNASeq at Day 2 timepoints
Time Frame: Day 2 (48 hr post feeding)
Reporting Status: Not Posted, anticipated posting 2022-12

3. Secondary Outcome: Flow Cytometry Analysis of PBMCs Collected Day 0 (Baseline) and Days 2 and 14 After Feeding for Saliva-specific T-cells
Description: Describing and understanding cellular immunity to Aedes saliva in heavily exposed individuals will simulate endemic conditions and will inform vaccine design in these target populations.
Time Frame: Day 14
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Two weeks
Description: Adverse events were collected according to definition of adverse events by clinicaltrials.gov
Arm/Group | Mosquito Feeding
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT04350905/Prot_SAP_000.pdf